CLINICAL TRIAL: NCT05506592
Title: Evaluation of the Efficacy of an Anti Dandruff Shampoo Against Placebo on Dandruff and Scalp Microflora Composition After 4 Weeks of Treatment and 4 Weeks of Relapse
Brief Title: Evaluation of the Efficacy of SeS2 Shampoo on Subjects Having Dandruff
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: L'Oreal (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACR_VICO_1411
Record Dates: First submitted 2022-08-12; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Dandruff
Keywords: Squamous; Malassezia; bacteria
MeSH Terms: conditions — Dandruff

STUDY DESIGN:
Intervention Model Description: To evaluate the impact of an anti-dandruff shampoo compared to vehicle (placebo) on scalp microflora composition after 4 weeks of treatment and 4 weeks of relapse, on healthy volunteers with moderate to severe dandruff status
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selenium disulfide shampoo (Active Comparator)
  Interventions: Other: dermatological product
- placebo shampoo (Placebo Comparator)
  Interventions: Other: dermatological product

INTERVENTIONS:
Other: dermatological product — cosmetic shampoo

SUMMARY:
A shampoo containing SeS2 was evaluated versus placebo on healthy subjects suffering from dandruff in order to assess clinical benefits and its impact on fungal and bacterial scalp microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers;
2. Age: 18 to 60 years old included;
3. Phototype (Fitzpatrick): I to IV;
4. Subjects with hair length > 2 cm, and preferentially shorter than shoulder length;
5. Females of childbearing potential, who are sexually actives, using an effective contraceptive method* for at least one month before the beginning of the study, and throughout the study;
6. Subjects exhibiting moderate to severe dandruff status of scalp at screening
7. Subjects having at inclusion visit Day 0:
8. total dandruff score (adherent + non-adherent) > or = 4.5 (ranging from 0 to 10);
9. adherent dandruff score > or = 2.5 (ranging from 0 to 5);
10. no limit for non-adherent dandruff score;
11. Subjects having on inclusion Day 0, 2 areas with dandruff (score > 2.5) (one of 1x1cm2, the other of 2 x 2cm2) and 2 areas without dandruff (score < 1) (one of 1x1cm2, the other of 2 x 2cm2) in the vertex if possible
12. Subjects usually using a shampoo 3 times/week and willing to have three times/week shampoos during the course of the study;
13. Subjects agreeing to use only the supplied shampoo during all the study;
14. Subjects agreeing to have 4 hair areas on the scalp (2 areas of approximately 2 cm x 2 cm and 2 areas approximately 1cmx1cm) for micro flora sample taking (swabs);
15. Subjects agreeing to have hair cut around the 4 identified areas (zone of 1x0.5cm cut on the high corner of each area sampling)
16. Subjects who demonstrate understanding of the study and willingness to participate as evidenced by voluntary written informed consent and have received a signed and dated copy of the informed consent form.
17. Subject affiliated to a social security or insurance system;
18. Subjects willing to comply to the study requirements;
19. Subjects who are willing not to take part in another clinical study in another investigating centre;
20. Subjects who agree to give accurate personal information;
21. Subjects who are able to attend all study visits. * The effective contraceptive methods: sexually active females of childbearing potential should either be surgically sterile (oophorectomy, hysterectomy or tubal ligation), or should use a medically accepted contraceptive regimen: systemic contraceptive (oral, implant, injection), diaphragm or cervical cap with intravaginal spermicide,intravaginal device, intrauterine device (IUD), condom with spermicide

Exclusion Criteria:

Inclusion Criteria

1. Healthy male or female volunteers;
2. Age: 18 to 60 years old included;
3. Phototype (Fitzpatrick): I to IV;
4. Subjects with hair length > 2 cm, and preferentially shorter than shoulder length;
5. Females of childbearing potential, who are sexually actives, using an effective contraceptive method* for at least one month before the beginning of the study, and throughout the study;
6. Subjects exhibiting moderate to severe dandruff status of scalp at screening and at D-3;
7. Subjects having at inclusion visit Day 0:
8. total dandruff score (adherent + non-adherent) > or = 4.5 (ranging from 0 to 10);
9. adherent dandruff score > or = 2.5 (ranging from 0 to 5);
10. no limit for non-adherent dandruff score;
11. Subjects having on inclusion Day 0, 2 areas with dandruff (score > 2.5) (one of 1x1cm2, the other of 2 x 2cm2) and 2 areas without dandruff (score < 1) (one of 1x1cm2, the other of 2 x 2cm2) in the vertex if possible
12. Subjects usually using a shampoo 3 times/week and willing to have three times/week shampoos during the course of the study;
13. Subjects agreeing to use only the supplied shampoo during all the study;
14. Subjects agreeing to have 4 hair areas on the scalp (2 areas of approximately 2 cm x 2 cm and 2 areas approximately 1cmx1cm) for micro flora sample taking (swabs);
15. Subjects agreeing to have hair cut around the 4 identified areas (zone of 1x0.5cm cut on the high corner of each area sampling)
16. Subjects who demonstrate understanding of the study and willingness to participate as evidenced by voluntary written informed consent and have received a signed and dated copy of the informed consent form.
17. Subject affiliated to a social security or insurance system;
18. Subjects willing to comply to the study requirements;
19. Subjects who are willing not to take part in another clinical study in another investigating centre;
20. Subjects who agree to give accurate personal information;
21. Subjects who are able to attend all study visits. * The effective contraceptive methods: sexually active females of childbearing potential should either be surgically sterile (oophorectomy, hysterectomy or tubal ligation), or should use a medically accepted contraceptive regimen: systemic contraceptive (oral, implant, injection), diaphragm or cervical cap with intravaginal spermicide,intravaginal device, intrauterine device (IUD), condom with spermicide

Exclusion Criteria

1. Subjects with any systemic disorder or skin disease that would, in the investigator's judgment, significantly affect the interpretation of the study results (e.g. seborrheic dermatitis which shows the syndrome of invasion plaque and/or pityriasis amiantacea, atopic dermatitis, eczema or psoriasis);
2. Subjects with cutaneous affection of the scalp (psoriasis, atopic dermatitis, seborrheic dermatitis which shows the syndrome of invasion plaque and/or pityriasis amiantacea, …);
3. Female subjects who are known to be pregnant or who are intending to become pregnant over the duration of the study;
4. Female subjects who are currently breast-feeding or have been breast-feeding in the 6 months prior to the start of the study;
5. Male subjects with alopecia grade ≥ V according to Hamilton-Norwood patterns, female subjects with alopecia grade I, II or III according to Ludwig patterns;
6. Subjects with frizzy hair influencing the scoring of dandruff;
7. Subjects with significant white hair influencing the scoring of dandruff;
8. Subjects who have skin marks on the scalp that could interfere with the assessments (e.g. pigmentation, tattoo, scarring etc.);
9. Subjects who have used products for the scalp (dyeing, bleaching, permanent waving and straightening …) within the three weeks prior to the study;
10. Subjects who have used anti-dandruff treatment (per os or topical) during the last three weeks before the start of the study;
11. Subjects who have used cosmetic anti-hairloss treatment (per os or topical) during the last three months before the start of the study, or/and subject who has used medical anti-hair loss treatment (per os or topical, ex: Minoxidil, finasteride, etc…) during the last six months before the start of the study;
12. Subjects with personal history of allergy and/or particular reactivity to antidandruff products, and/or to cosmetic products containing tensioactive agents (soaps, shower gel, conditioner …), and/or to latex;
13. Subjects who have taken any systemic drug containing corticoids, or anti-fungal, or antibiotics, or any prolonged use of topical drug containing corticoids, or anti-fungal, or antibiotics, or any prolonged use of non-steroidal anti-inflammatory, or anti-histaminic within one month prior to the study;
14. Subjects who have taken retinoic acid since less than three months prior to the study;
15. Subjects receiving other medication which, in the opinion of the investigator, will affect either the scientific validity of the study or the subject's wellbeing.
16. Subjects with a history of medical/surgical events (or surgical events planned) which, in the opinion of the investigator, will affect either the scientific validity of the study or the subject's wellbeing;
17. Immunosuppressed subject;
18. Subjects with medical history of skin cancer;
19. Subjects who have started, stopped or changed his/her hormonal treatment (including contraceptive pill) in the previous one month prior to the study;
20. Subjects practicing regularly water sports and/or having regularly sauna sessions;
21. Subjects exposed to the sun or UV rays in an excessive way during the last month prior to the study (according to the investigator);
22. Subjects deprived of liberty by adjunction or by official decision;
23. Subjects who are participating or who has participated to a clinical study for which the exclusion period is not finished;
24. Subjects unable to be contacted by phone;
25. Subjects belonging to the staff of the investigating centre

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Analysis of microflora from swabs for fungi quantification | 1 month
  malassezia qPCR
Analysis of microflora from swabs for bacteria quantification | 1 month
  Cutibacterium qPCR
Analysis of microflora from swabs for bacteria diversity | 1 month
  sequencing 16S
Analysis of microflora from swabs for fungi diversity | 1 month
  sequencing ITS

SECONDARY OUTCOMES:
Grading of Dandruff severity | 1 month
  Dandruff severity 0-5 ordinal scale

OTHER OUTCOMES:
Clinical assessment of oily aspect of the scalp | 1 month
  oily aspect of the scalp 1-5 ordinal scale
Clinical assessment of erythema | 1 month
  erythema 0-5 ordinal scale
Self-perception of efficacy: dandruff | 1 month
  Self-perception of dandruff 5-point-scale
Self-perception of efficacy greasy aspect | 1 month
  Self-perception of greasy 10-point-scale
Self-perception of efficacy global efficacy | 1 month
  Self-perception of global efficacy 5-point-scale

CONTACTS AND LOCATIONS:
Locations (1):
- Interteck, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided